CLINICAL TRIAL: NCT01859962
Title: A Phase 2a Study of PPI-668 in Combination With BI 207127 and Faldaprevir, With and Without Ribavirin, in Treatment-Naive Patients With Chronic Hepatitis C (HCV Genotype 1a)
Brief Title: Study of PPI-668, BI 207127 and Faldaprevir, With and Without Ribavirin, in the Treatment of Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Presidio Pharmaceuticals, Inc. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPI-668-201
Record Dates: First submitted 2013-05-17; First posted 2013-05-22 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Hepatitis C
Keywords: Liver diseases; Virus diseases; Ribavirin; protease inhibitor; NS5B polymerase inhibitor; NS5A inhibitor
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Diseases; Virus Diseases | interventions — ravidasvir; faldaprevir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PPI-668, BI 207127 Dose 1, Faldaprevir, and Ribavirin (Active Comparator): PPI-668, BI 207127 Dose 1, Faldaprevir, and Ribavirin dosed in combination
  Interventions: Drug: PPI-668; Drug: BI 207127 Dose 1; Drug: Faldaprevir; Drug: Ribavirin
- PPI-668, BI 207127 Dose 2, Faldaprevir, and Ribavirin (Active Comparator): PPI-668, BI 207127 Dose 2, BI 207127 Placebo, Faldaprevir, and Ribavirin dosed in combination
  Interventions: Drug: PPI-668; Drug: BI 207127 Dose 2; Drug: Faldaprevir; Drug: Ribavirin; Drug: BI 207127 Placebo
- PPI-668, BI 207127 Dose 1, and Faldaprevir (Active Comparator): PPI-668, BI 207127 Dose 1, and Faldaprevir dosed in combination
  Interventions: Drug: PPI-668; Drug: BI 207127 Dose 1; Drug: Faldaprevir

INTERVENTIONS:
Drug: PPI-668
Drug: BI 207127 Dose 1
  Arms: PPI-668, BI 207127 Dose 1, Faldaprevir, and Ribavirin; PPI-668, BI 207127 Dose 1, and Faldaprevir
Drug: BI 207127 Dose 2
  Arms: PPI-668, BI 207127 Dose 2, Faldaprevir, and Ribavirin
Drug: Faldaprevir
Drug: Ribavirin
  Arms: PPI-668, BI 207127 Dose 1, Faldaprevir, and Ribavirin; PPI-668, BI 207127 Dose 2, Faldaprevir, and Ribavirin
Drug: BI 207127 Placebo
  Arms: PPI-668, BI 207127 Dose 2, Faldaprevir, and Ribavirin

SUMMARY:
This study is designed to provide a preliminary assessment of the safety and effectiveness of the combination of PPI-668, BI 207127 and faldaprevir, with or without ribavirin, in the treatment of chronic hepatitis C virus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 65 years of age; if females are of childbearing potential, then they must be willing to use two non-hormonal methods of birth control
2. Body weight greater than 40 kg and less than 125 kg
3. Clinical diagnosis of chronic hepatitis C
4. Treatment-naïve for hepatitis C: no previous treatment with interferon, pegylated interferon, ribavirin, telaprevir, boceprevir, or any investigational therapies for hepatitis C
5. No symptoms or signs of intercurrent illness at Screen (other than those attributable to hepatitis C)
6. No clinically significant abnormalities in the 12-lead electrocardiogram at Screen
7. Signed informed consent prior to trial participation.

Exclusion Criteria:

1. Seropositive for HIV antibody or Hepatitis B Surface Antigen at Screen
2. Liver disease due to causes other than chronic HCV infection
3. Symptoms or signs of decompensated liver disease, or evidence of cirrhosis
4. Any medical condition that may interfere with the absorption, distribution or elimination of study drugs
5. Poorly controlled or unstable hypertension at Screen.
6. Clinically significant, unstable cardiovascular or pulmonary disease, including cardiovascular or pulmonary disease requiring pharmacologic intervention other than anti-hypertensive medications, statins, and/or prophylactic aspirin (or similar anticoagulant).
7. Red blood cell disorder, including (but not limited to): thalassemia major or minor, sickle cell anemia.
8. Diabetes Mellitus treated with insulin or hypoglycemic agents
9. History of asthma requiring hospital admission within the preceding 12 months
10. History of alcohol abuse or illicit drug use which could interfere with a patient's compliance with the protocol requirements, or with the safety or efficacy assessments in this study
11. Patients requiring treatment, during this study, with any of the medications on the restricted medications list (provided in the investigator site file), are not eligible for this study due to considerations of possible drug interactions with the study drug regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients achieving sustained viral response (SVR) | 12 weeks after the end of treatment

SECONDARY OUTCOMES:
Proportion of patients with "virologic relapse" post-treatment, defined as confirmed and quantifiable (>LLOQ) serum HCV RNA in a patient who achieved non-detectable serum HCV RNA by the end of treatment | up to 24 weeks post-treatment
Proportion of patients with confirmed viral breakthrough during study treatment | up to 12 weeks of study treatment
  "Confirmed viral breakthrough" is defined as a > 1 log increase in HCV RNA from post-Baseline nadir value or confirmed increase in HCV RNA ≥LLOQ if HCV RNA previously declined to <LLOQ (detected or not detected), during the 12-week study treatment period
Proportions of study participants who receive at least one dose of study drug and who prematurely discontinue study treatment, and proportions prematurely discontinuing treatment for clinical adverse events or laboratory abnormalities | up to 12 weeks of study treatment
Proportions of study participants experiencing treatment-emergent adverse events (serious and non-serious) considered to be possibly or probably attributable to study treatment, overall and by body system | up to 12 weeks of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Brown, MD, Study Director — Presidio Pharmaceuticals, Inc.
Locations (1):
- Quest Clinical Research, San Francisco, California, United States